CLINICAL TRIAL: NCT05894174
Title: The Effect of Board Game-Based Nutrition Education on Primary School Children's Nutrition Behaviors, Self-Efficacy and Attitudes
Brief Title: The Effect of Board Game-Based Nutrition Education on Primary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Kent University (Other)
Responsible Party: Principal Investigator, Beyzanur Çamlıbel, Research Assistant, Istanbul Kent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KENT-BES-BC-01
Record Dates: First submitted 2023-05-18; First posted 2023-06-08 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Nutrition Assessment; Education; Child Behavior
Keywords: Dietary Intake; Behavior; Self Efficacy; Attitude
MeSH Terms: conditions — Child Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: Two groups with the intervention group in which the game was applied and the control group
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be performed by a investigator who was blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group refers to the group that will the "Food Hunter" board game intervention developed by the researchers to enable children to recognize healthy and unhealthy foods; to learn what vitamins and minerals are necessary for children in the growth and development period, their effects on our health and in which foods they are found.
  Interventions: Behavioral: Board Game
- Control Group (No Intervention): The control group refers to the group that will not receive any nutrition education intervention.

INTERVENTIONS:
Behavioral: Board Game — Food Hunter board game intervention, which includes various nutrient cards and question cards and is played with pawns and dice, will be played with children for approximately 4 weeks, one day a week and one session (40 minutes) with the researcher dietitian. By talking about the nutrients in the game on the game cards, children will be able to recognize the nutrients and important points will be emphasized for the participants with the answers to the cards containing various questions about healthy nutrition.
  Arms: Intervention Group

SUMMARY:
The purpose of this study to design a board game that will enable primary school children to recognize foods by enabling them to distinguish between healthy and unhealthy foods by going beyond the traditional education patterns and to compare the effects of this board game-based nutrition education intervention on children's behaviors, self-efficacy, and attitudes with the control group in which no intervention was made.

DETAILED DESCRIPTION:
Nutrition is an important part of health and development. In particular, the gaining of healthy eating habits in early childhood promotes growth and development and reduces the risk of many non-communicable diseases, especially obesity. In order to create healthy societies in the future, nutrition education is one of the effective methods for developing healthy eating behaviors and raising awareness starting from childhood. Game-based education approaches provide motivation for learning information that is made a part of the game by going beyond traditional education methods. Board games are used in nutrition education by giving children the opportunity to think interactively and make different choices with their immersive stories and designs.

ELIGIBILITY:
Inclusion Criteria:

* In the 3 schools where the study will be carried out
* 4th grade student
* Does not have any physical disability related to vision, hearing and speech
* Without any chronic or metabolic disease

Exclusion Criteria:

* Having any chronic or metabolic disease
* Can't read and write

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Food Behavior Scale (FBS) | Baseline and four weeks
  It was developed to measure children's habit of consuming low-fat/salt foods in contrast to high-fat/salt food options. A validity and reliability study was conducted (Cronbach's alpha coefficient 0.68). The items of the scale consisting of 14 questions with 2 options take a value of -1 for unhealthy food and +1 for healthy food and the total score varies between -14 and +14. A high total score on the scale indicates healthy eating habits.
Change in Children's Dietary Self- Efficacy Scale (CDSS) | Baseline and four weeks
  It was developed to measure children's self-confidence to choose low-fat and low-salt foods despite the fatty and salty food options. A reliability and validity study was conducted (Cronbach's alpha coefficient 0.79). It is a 3-point Likert-type scale consisting of 15 items. Scale items can be scored between -1 and +1 (-1: not sure, 0: somewhat sure, +1: very sure) and the total score varies between -15 and +15. A high total score on the scale indicates a high self-efficacy value.
Change in Nutrition Attitude Subscale (NAS) | Baseline and four weeks
  It's the nutrition-related subscale of the Child Heart Health Promotion Attitude Scale, which normally consists of 4 subscales with 16 questions. The aim of the scale is to assess the heart health promotion attitudes of school-age children. The validity and reliability of this Likert-type scale has been studied (Cronbach's alpha coefficient 0.68). In the study, the scale consists of 4 questions and the scale items are scored as 1 "strongly disagree" and 4 "strongly agree" and the total score that can be obtained varies between a minimum of 4 and a maximum of 16 points. A high total score indicates a positive attitude.

SECONDARY OUTCOMES:
Change in The Food Frequency Questionnaire (FFQ) | Baseline and four weeks
  It is a food consumption frequency form with 16 nutrients. Participants were required to indicate the frequency of consumption of the specified foods and meals by selecting one of the following options: "every day (5), 5-6 days a week (4), 3-4 days a week (3), 1-2 days a week (2), 1-2 days a month (1) and never (0)".

CONTACTS AND LOCATIONS:
Overall Officials: Beyzanur Çamlıbel, Principal Investigator — Istanbul Kent University
Locations (1):
- Beyzanur Çamlıbel, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No